CLINICAL TRIAL: NCT07079124
Title: A Multilevel Social Participation Intervention for Older Adults in Nursing Homes: Development and Implementation Based on the Social Ecological Model
Brief Title: Social Participation Program for Older Adults in Nursing Homes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Huang Chenshan, MD, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025[302]
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Older Adults
Keywords: older adults; social participation; nursing home; cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Participation Intervention (Experimental): Participants in this group will receive a 12-week multi-level social participation intervention based on the Social Ecological Model. The intervention includes individual-level goal setting, interpersonal-level group activities, and organizational-level environmental support. Intervention components consist of a health education manual, activity and social resource toolkit, motivational participation package, and staff training sessions. Activities are conducted twice per week.
  Interventions: Behavioral: Multi-level Social Participation Intervention
- Health Education (Active Comparator): Participants in the health education group will receive standardized health education materials during the 12-week study period, without participating in the structured multi-level social participation intervention. After study completion, they will be offered the opportunity to join the full intervention program if they wish.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Multi-level Social Participation Intervention — The intervention will span 12 weeks and comprises five core components: (1) a health education manual, (2) a resource information package, (3) a structured library of social activities, (4) a motivational incentive kit, and (5) a training toolkit for staff.
  Arms: Social Participation Intervention
Behavioral: Health Education — Standardized Health Education Materials
  Arms: Health Education

SUMMARY:
The goal of this clinical trial is to learn whether a multi-level social participation program can help improve social engagement and slow down cognitive decline in older adults living in nursing homes. The main questions it aims to answer are:

Can this program improve how often and how meaningfully participants engage in social activities?

Can this program help maintain or improve participants' cognitive abilities?

Researchers will compare this program to a health education group to see if it is more effective in supporting social participation and cognitive health.

Participants will:

Join a 12-week program that includes group activities, personalized support, staff assistance, and health education content

Be assessed before and after the program using cognitive and social participation questionnaires

Be randomly assigned to either the multi-level social participation program group or the health education group

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility and effectiveness of a multi-level social participation intervention among older adults residing in nursing homes, based on the Social Ecological Model (SEM). Against the backdrop of accelerated aging and rising dementia prevalence in institutional settings, the intervention seeks to enhance social engagement and mitigate cognitive decline through a structured, multi-dimensional approach.

A total of 120 older adults aged 60 years and above will be recruited from nursing homes and randomly assigned to either the intervention group or a health education group. The intervention will span 12 weeks and comprises five core components:

1. a health education manual,
2. a resource information package,
3. a structured library of social activities,
4. a motivational incentive kit, and
5. a training toolkit for staff.

The intervention addresses three levels of influence:

1. Individual level: enhancing motivation and cognitive engagement through behavior activation strategies;
2. Interpersonal level: fostering peer interaction and support networks;
3. Organizational level: enabling supportive environments through staff training and institutional support.

Assessments will be conducted at baseline and post-intervention. The health education group will receive standardized health education materials during the study. This trial will provide empirical evidence for a scalable model of dementia prevention through social participation in institutional settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Basic comprehension and verbal communication abilities
* Resided in a long-term care facility for at least one month

Exclusion Criteria:

* Clinically diagnosed with dementia (based on DSM-IV-R criteria)
* Presence of severe physical illness or psychiatric disorder
* Significant visual or hearing impairments that may interfere with accurate cognitive assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive function assessed by the Montreal Cognitive Assessment (MoCA) | From enrollment to the end of treatment at 12 weeks.
  The Montreal Cognitive Assessment (MoCA) will be used to assess global cognitive function, including attention, memory, language, visuospatial skills, and executive functions, with scores ranging from 0 to 30, where higher scores indicate better cognitive performance.

SECONDARY OUTCOMES:
Social participation | At baseline and the end of treatment at 12 weeks.
  Social participation will be measured through four instruments:
  1. The Social Support Rating Scale (SSRS) (12-66 points; higher scores indicate better social support);
  2. Lubben Social Network Scale-6 (LSNS-6) (0-30 points; higher scores indicate stronger social networks);
  3. Community Participation Index (CPI) (0-113 points; higher scores indicate more frequent social engagement);
  4. The interRAI LTCF Social Participation Index (0-6 points; higher scores indicate greater social involvement).
Loneliness | At baseline and the end of treatment at 12 weeks.
  The 8-item UCLA Loneliness Scale (ULS-8) will be used (8-32 points; higher scores indicate greater loneliness).
Change in health-related quality of life (HRQoL) assessed by EQ-5D-5L | From enrollment to the end of treatment at 12 weeks.
  The EQ-5D-5L will be used, including: Utility index (higher scores indicate better health); Visual analog scale (0-100; higher scores indicate better health)
Psychological state | At baseline and the end of treatment at 12 weeks.
  1. Geriatric Depression Scale-15 (GDS-15) (0-15 points; higher scores indicate more severe depression);
  2. Self-Rating Anxiety Scale (SAS) (25-100 standard score; higher scores indicate more severe anxiety).
Cost-benefit | At the end of treatment at 12 weeks.
  The EQ-5D-5L questionnaire will be used to calculate quality-adjusted life years for cost-effectiveness analysis.
Fidelity | At the end of treatment at 12 weeks.
  Intervention fidelity checklist
Compliance | At the end of treatment at 12 weeks.
  Attendance rate
Intervention satisfaction with intervention measured by 5-point Likert scale | At the end of treatment at 12 weeks.
  The Intervention Satisfaction Evaluation Questionnaire (self-developed) will be used (9-45 points; higher scores indicate greater satisfaction with the intervention).
Incidence of intervention-related adverse events (AEs) recorded by Self-compiled questionnaire | At the end of treatment at 12 weeks.
  Intervention-related adverse event record form
Intervention acceptability | At the end of treatment at 12 weeks.
  The Intervention Acceptability Assessment Scale (based on the Theory of Acceptance and Use of Technology framework) will be used (8-40 points; higher scores indicate greater acceptability of the intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No